CLINICAL TRIAL: NCT06367465
Title: Feasibility and Acceptability of Early Linkage to HCV Treatment in Pregnancy Feasibility and Acceptability of Early Linkage to HCV Treatment in Pregnancy
Brief Title: Feasibility and Acceptability of HCV Treatment in Pregnancy
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 202308056
Record Dates: First submitted 2024-03-06; First posted 2024-04-16 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis C; Pregnancy Complications
MeSH Terms: conditions — Hepatitis C; Pregnancy Complications | interventions — glecaprevir and pibrentasvir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Female patients ≥ 18 years old, pregnant at the time of study intake, diagnosed with hepatitis c: Female patients ≥ 18 years old, pregnant at the time of study intake, diagnosed with hepatitis c virus infection and a history of past or current drug use.
  Interventions: Drug: Glecaprevir-pibrentasvir

INTERVENTIONS:
Drug: Glecaprevir-pibrentasvir — Glecaprevir-pibrentasvir 100 mg / 40 mg 3 tab orally (PO) once daily for 56 days.

SUMMARY:
Pregnant adults over the age of 18 who are seen in the Washington University obstetrics and gynecology, maternal fetal medicine or infectious diseases clinic or admitted to BJH with hepatitis C virus infection who have a history of past or current drug use

Participant Duration: Approximately 1 year.

Aims:

Aim 1 - Evaluate adherence and treatment completion rates when glecaprevir-pibrentasvir is started during pregnancy for women who use drugs.

Aim 2 - Evaluate patient experience with hepatitis C virus treatment during pregnancy.

DETAILED DESCRIPTION:
Pregnant adults over the age of 18 with a history of either past or current drug use who are seen in the Washington University obstetrics and gynecology, maternal fetal medicine or infectious diseases clinic or admitted to BJH with hepatitis C virus infection who consent to participate in the study will be treated with glecaprevir-pibrentasvir.

All consented individuals will participate in four (4) in-person study visits. At the first in-person study visit, patients will receive information about hepatitis C virus treatment, complete testing for HIV and HBV and be assessed for cirrhosis. Patients who meet study criteria will initiate HCV treatment with glecaprevir-pibrentasvir. Patients will return for a second in-person study visit while on HCV treatment (between day 14-56) at which time they will complete a questionnaire about medication adherence and have HCV RNA testing performed. A third in-person study visit will occur at completion of HCV treatment at which time patients will again complete a questionnaire about medication adherence, and have HCV RNA testing performed. The final study visit will occur 4 weeks after completion of HCV treatment at which time patients will have HCV RNA testing performed. All labs that are included as part of the study are standard of care labs for all pregnant women, and are standard of care during HCV treatment (HCV RNA, CBC and CMP).

Additional information about the clinical course of infection (including HCV RNA testing obtained at the time of labor and delivery), and maternal and fetal outcomes will be abstracted from the medical record at 1 year post study enrollment.

All participants will be followed longitudinally in the medical record to ascertain maternal and fetal outcomes and HCV re-infections for up to 1 year post study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥ 18 years old, pregnant at the time of study intake, diagnosed with hepatitis c virus infection and a history of past or current drug use.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Adults over the age of 18 with hepatitis C virus infection who are currently pregnant with a history of past or current drug use. Patients must have health insurance which covers hepatitis C virus treatment with direct acting antivirals and who agree to begin HCV treatment with glecaprevir-pibrentasvir during pregnancy. Participants pregnancies must have reached at least 10 weeks gestational age prior to initiation of medication. Adults over the age of 18 with hepatitis C virus infection who are currently pregnant with a history of past or current drug use. Patients must have health insurance which covers hepatitis C virus treatment with direct acting antivirals and who agree to begin HCV treatment with glecaprevir-pibrentasvir during pregnancy. Participants pregnancies must have reached at least 10 weeks gestational age prior to initiation of medication.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Medication adherence and treatment completion rates. | 2 years
  The primary objective of this study is to assess patient adherence and treatment completion rates of women with a history of past or current drug use who receive initiation of Hepatitis C Virus treatment with glecaprevir-pibrentasvir during pregnancy. The primary objective of this study is to assess patient adherence and treatment completion rates of women with a history of past or current drug use who receive initiation of Hepatitis C Virus treatment with glecaprevir-pibrentasvir during pregnancy.

SECONDARY OUTCOMES:
Patient satisfaction Questionnaire | 2 years
  To assess patient satisfaction with early initiation of glecaprevir-pibrentasvir during pregnancy.
Virologic outcome and clinical success at Day 28 post treatment | 2 years
  Virologic and clinical outcomes at 4 weeks after completion of glecaprevir-pibrentasvir between patients who received glecaprevir-pibrentasvir during pregnancy and to those who received it post-partum.
Sample size estimation for future study | 2 years
  Sample size estimation for future study

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Barnes Jewish Hospital, St Louis, Missouri
  - Washington Univeristy, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossi RM, Wolfe C, Brokamp R, McAllister JM, Wexelblatt S, Warshak CR, Hall ES. Reported Prevalence of Maternal Hepatitis C Virus Infection in the United States. Obstet Gynecol. 2020 Feb;135(2):387-395. doi: 10.1097/AOG.0000000000003644. PMID 31923064
- [Background] ACOG Committee Opinion No. 736: Optimizing Postpartum Care. Obstet Gynecol. 2018 May;131(5):e140-e150. doi: 10.1097/AOG.0000000000002633. PMID 29683911
- [Background] Bryant AS, Haas JS, McElrath TF, McCormick MC. Predictors of compliance with the postpartum visit among women living in healthy start project areas. Matern Child Health J. 2006 Nov;10(6):511-6. doi: 10.1007/s10995-006-0128-5. PMID 16807794
- [Background] Wilcox A, Levi EE, Garrett JM. Predictors of Non-Attendance to the Postpartum Follow-up Visit. Matern Child Health J. 2016 Nov;20(Suppl 1):22-27. doi: 10.1007/s10995-016-2184-9. PMID 27562797
- [Background] Weir S, Posner HE, Zhang J, Willis G, Baxter JD, Clark RE. Predictors of prenatal and postpartum care adequacy in a medicaid managed care population. Womens Health Issues. 2011 Jul-Aug;21(4):277-85. doi: 10.1016/j.whi.2011.03.001. Epub 2011 May 12. PMID 21565526
- [Background] Bushman ET, Subramani L, Sanjanwala A, Dionne-Odom J, Franco R, Owen J, Subramaniam A. Pragmatic Experience with Risk-based versus Universal Hepatitis C Screening in Pregnancy: Detection of Infection and Postpartum Linkage to Care. Am J Perinatol. 2021 Sep;38(11):1109-1116. doi: 10.1055/s-0041-1728827. Epub 2021 May 2. PMID 33934324
- [Background] Jarlenski M, Chen Q, Ahrens KA, Allen L, Austin AE, Chappell C, Donohue JM, Hammerslag L, Lanier P, McDuffie MJ, Talbert J, Tang L, Krans EE; Medicaid Outcomes Distributed Research Network (MODRN). Postpartum Follow-up Care for Pregnant Persons With Opioid Use Disorder and Hepatitis C Virus Infection. Obstet Gynecol. 2022 May 1;139(5):916-918. doi: 10.1097/AOG.0000000000004760. Epub 2022 Apr 5. PMID 35576352
- [Background] Epstein RL, Sabharwal V, Wachman EM, Saia KA, Vellozzi C, Hariri S, Linas BP. Perinatal Transmission of Hepatitis C Virus: Defining the Cascade of Care. J Pediatr. 2018 Dec;203:34-40.e1. doi: 10.1016/j.jpeds.2018.07.006. Epub 2018 Aug 28. PMID 30170857
- [Background] Kushner T, Lange M, Sperling R, Dieterich D. Treatment of Women With Hepatitis C Diagnosed in Pregnancy: a Co-Located Treatment Approach. Gastroenterology. 2022 Nov;163(5):1454-1456.e1. doi: 10.1053/j.gastro.2022.07.017. Epub 2022 Jul 18. No abstract available. PMID 35863531
- [Background] Zeng QL, Yu ZJ, Lv J, Zhang HX, Wang B, Dong XP, Chen ZM, Cui GL, Ji F. Sofosbuvir-based therapy for late pregnant women and infants with severe chronic hepatitis C: A case series study. J Med Virol. 2022 Sep;94(9):4548-4553. doi: 10.1002/jmv.27877. Epub 2022 Jun 1. PMID 35595682
- [Background] AbdAllah M, Alboraie M, Abdel-Razek W, Hassany M, Ammar I, Kamal E, Alalfy M, Okasha A, El Akel W, Shaaban E, Elbaz T, Hefny Z, Gomaa A, El-Bendary M, El-Serafy M, Esmat G, Doss W, El-Sayed MH. Pregnancy outcome of anti-HCV direct-acting antivirals: Real-life data from an Egyptian cohort. Liver Int. 2021 Jul;41(7):1494-1497. doi: 10.1111/liv.14913. Epub 2021 May 11. PMID 33905164
- [Background] Chappell CA, Scarsi KK, Kirby BJ, Suri V, Gaggar A, Bogen DL, Macio IS, Meyn LA, Bunge KE, Krans EE, Hillier SL. Ledipasvir plus sofosbuvir in pregnant women with hepatitis C virus infection: a phase 1 pharmacokinetic study. Lancet Microbe. 2020 Sep;1(5):e200-e208. doi: 10.1016/S2666-5247(20)30062-8. Epub 2020 Jul 27. PMID 32939459
- [Background] Bhattacharya D, Aronsohn A, Price J, Lo Re V; AASLD-IDSA HCV Guidance Panel. Hepatitis C Guidance 2023 Update: AASLD-IDSA Recommendations for Testing, Managing, and Treating Hepatitis C Virus Infection. Clin Infect Dis. 2023 May 25:ciad319. doi: 10.1093/cid/ciad319. Online ahead of print. PMID 37229695